CLINICAL TRIAL: NCT00591552
Title: Use of Harmonic Scalpel to Decrease Lymphatic and Chest Tube Drainage After Lymph Node Dissection With Lobectomy. A Single Center Prospective Randomized Controlled Study.
Brief Title: Use of Harmonic Scalpel to Decrease Lymphatic and Chest Tube Drainage After Lymph Node Dissection With Lobectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sentara Cardiovascular Research Institute (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI-001; SCRI-001
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Lymph node dissection
MeSH Terms: conditions — Lung Neoplasms | interventions — Electrocoagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Electrocautery used for dissection.
  Interventions: Device: Electrocautery
- Group B (Active Comparator): Harmonic Scalpel used for dissection
  Interventions: Device: Harmonic ACE23P Scalpel

INTERVENTIONS:
Device: Harmonic ACE23P Scalpel — Lymph node dissection
  Arms: Group B
Device: Electrocautery
  Arms: Group A

SUMMARY:
In an effort to elucidate whether the Harmonic Scalpel will improve sealing lymphatics and decrease lymphatic drainage thereby decreasing the length of time that chest tubes are required and minimizing length of stay; the Harmonic Scalpel will be compared to a control group which uses electrocautery. This study will assess these two different methods to determine if there is a notable decrease in the amount of drainage with one versus the other.

DETAILED DESCRIPTION:
Lymph node dissection is an integral part of the surgical management of lung cancer. Knowledge of lymph node status plays a key role in therapeutic decision making and prognosis. Associated with this dissection comes the propensity for lymphatic leakage, increased chest tube drainage, prolonged retention of chest tubes in the postoperative period and increased patient length of stay. Our center performs complete mediastinal node dissection of all relevant regional lymph nodes which generally include paratracheal, pretracheal, subcarinal, hilar and paraesophageal nodes. The current standard of practice for the dissection of the lymph nodes includes the use of the Harmonic Scalpel or electrocautery. Known risk of electrocautery include localized nerve damage, cardiac arrhythmias and damage to the tissue sample/specimen that is used for pathology. The Harmonic Scalpel technology has recently become available for use. Current experience with the Harmonic Scalpel suggests that there is less localized nerve damage, less incidence of arrhythmias, less damage to the tissue sample and less lymph leakage. There is no published data to support this hypothesis, thus the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing resection for stage 1, 2 or 3A lung cancer.
* Patients between the ages of 20-75.

Exclusion Criteria:

* History of Congestive Heart Failure.
* History of renal failure, ie., creatinine greater than 2.2.
* Patients with bulky or matted lymph nodes in stage 3A.
* Current pregnancy.
* Current participation in another study involving an investigational device or drug.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-12; Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Amount of chest tube drainage | daily

SECONDARY OUTCOMES:
Pleural effusions monitored by chest x-ray. | Every other day and at four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Newton, MD, Principal Investigator — Sentara Cardiovascular Research Institute
Locations (1):
- Sentara Norfolk General Hospital/Sentara Heart Hospital, Norfolk, Virginia, United States

REFERENCES:
- [Background] Holub Z, Jabor A, Kliment L, Lukac J, Voracek J. Laparoscopic lymph node dissection using ultrasonically activated shears: comparison with electrosurgery. J Laparoendosc Adv Surg Tech A. 2002 Jun;12(3):175-80. doi: 10.1089/10926420260188065. PMID 12184902
- [Background] Lumachi F, Burelli P, Basso SM, Iacobone M, Ermani M. Usefulness of ultrasound scissors in reducing serous drainage after axillary dissection for breast cancer: a prospective randomized clinical study. Am Surg. 2004 Jan;70(1):80-4. PMID 14964555
- [Background] Kajiyama Y, Iwanuma Y, Tomita N, Amano T, Hattori K, Tsurumaru M. Sealing the thoracic duct with ultrasonic coagulating shears. Hepatogastroenterology. 2005 Jul-Aug;52(64):1053-6. PMID 16001628